CLINICAL TRIAL: NCT07155499
Title: A Two-stage Clinical Trial With Dose Escalation at the First Stage and a Single-blind, Placebo-controlled Clinical Trial for Evaluation of Efficacy, Safety, Reactogenicity and Immunogenicity of GNR-127 at the Second Stage in Patients With Allergic Rhinitis Sensitized to Birch Pollen.
Brief Title: A Clinical Trial for Evaluation of Efficacy, Safety and Immunogenicity of GNR-127 (Recombinant ABP Antigen Protein Which Carries a Birch Pollen Allergen [BET V 1] and an Apple Allergen [MAL D 1]) in Patients With Birch Pollen Allergic Rhinitis.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GNR127-BET01
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Hypersensitivity; Birch Pollen Allergy; Seasonal Allergy; Birch Pollen; Immune System Diseases; Respiratory Tract Diseases; Respiratory Hypersensitivity
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Immune System Diseases; Respiratory Tract Diseases; Respiratory Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Sequential - for first stage Parallel - for second stage
Who Masked: Participant, Investigator
Masking Description: Participant - for the second stage None (open label) - for the first stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GNR-127, 20 mcg (Experimental): GNR-127, 20 mcg, suspension for subcutaneous administration, 0.5 ml / dose
  Interventions: Biological: GNR-127, 20 mcg
- GNR-127, 40 mcg (Experimental): GNR-127 40 mcg, suspension for subcutaneous administration, 0.5 ml / dose
  Interventions: Biological: GNR-127, 40 mcg
- GNR-127, 80 mcg (Experimental): GNR-127 80 mcg, suspension for subcutaneous administration, 0.5 ml / dose
  Interventions: Biological: GNR-127, 80 mcg
- Placebo (Placebo Comparator): Suspension for subcutaneous administration, 0.5 ml / dose
  Interventions: Biological: GNR-127 placebo

INTERVENTIONS:
Biological: GNR-127, 20 mcg — GNR-127, 20 mcg in 0.5 ml administered 5 times every 4 weeks
  Other Names: Recombinant antigen protein carries a birch pollen allergen [BET V 1]
  Arms: GNR-127, 20 mcg
Biological: GNR-127, 40 mcg — GNR-127, 40 mcg in 0.5 ml administered 5 times every 4 weeks
  Other Names: Recombinant antigen protein carries a birch pollen allergen [BET V 1]
  Arms: GNR-127, 40 mcg
Biological: GNR-127, 80 mcg — GNR-127, 80 mcg in 0.5 ml administered 5 times every 4 weeks
  Other Names: Recombinant antigen protein carries a birch pollen allergen [BET V 1]
  Arms: GNR-127, 80 mcg
Biological: GNR-127 placebo — GNR-127 placebo 0.5 ml administered 5 times every 4 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is first-in-human phase 1/2 clinical trial to evaluate the safety, systemic and local reactogenicity of GNR-127 at the first stage in sequential cohorts of patients with allergic rhinitis with sensitization to the birch pollen, and then to determine and evaluate an effective and safe dose of the GNR-127 after five monthly administrations compared to placebo at the second stage.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is the most common disease in both children and adults and is a global health problem that affects approximately 400 million people worldwide. AR has a significant impact on the quality of life of patients, disrupting their sleep, physical and social activity.

AR is a disease characterized by IgE-mediated inflammation of the nasal mucosa (which develops under the influence of allergens) and the presence of at least two of the following symptoms that occur daily for an hour or more: nasal congestion (obstruction), nasal discharge (rhinorrhea), sneezing, itching in the nasal cavity. AR is often combined with other allergic diseases, such as allergic conjunctivitis, atopic dermatitis, and bronchial asthma.

The investigational product GNR-127 is a recombinant vaccine containing the ABP antigen protein, which includes the hypoallergenic peptides Bet v 1 (major birch allergen) and Mal d 1 (apple allergen), as well as the PreS protein of the hepatitis B virus as an immunogenic carrier. The drug is intended for the prevention of allergy to birch pollen - subcutaneous allergen immunotherapy (AIT) in patients suffering from AR with sensitization to birch pollen.

This study is a 'first-in-human' clinical trial and is aimed at evaluating the safety, systemic and local reactogenicity, preliminary efficacy and immunogenicity after the use of GNR-127.

This study is a two-stage study that combines phase I (Stage 1) and phase II (Stage 2) of a clinical trial.

Stage 1 (Phase I) is an open-label safety study of increasing doses of the investigational drug GNR-127 in patients with AR with sensitization to birch pollen.

Phase 1 is to evaluate the safety of three doses of GNR-127 and to determine the dose(s) to be studied in Phase 2. Patients enrolled in Phase 1 will continue to participate in the study in the appropriate dose cohort or prematurely complete their participation in the clinical study.

Phase 2 (Phase II) to be conducted as a single-blind, randomized, placebo-controlled trial. The main goal of Stage 2 is to determine the effective and safe dose of the investigational product in patients with AR with sensitization to birch pollen.

ELIGIBILITY:
Inclusion Criteria:

1. Having written informed consent to participate in the study obtained from the patient prior to the start of any procedures related to the study.
2. Men and women aged 18-55 years at the time of signing the informed consent.
3. Documented allergic rhinitis (AR) with a history of sensitization to birch pollen for at least 2 years prior to signing an informed consent.
4. Body mass index (BMI) 18.5≤BMI≤29.9 kg / m2.
5. Positive skin test (pric test) for the birch pollen allergen papule (blister) ≥ 3 mm at Screening.
6. A positive result for the presence of specific IgE to birch pollen in blood serum (sensitization level of class 2 and higher, which corresponds to quantitative indicators ≥ 0.7 kU/l) at Screening.
7. Consent to use a reliable method of contraception in accordance with the clinical trial protocol for the entire duration of participation in the study.

Exclusion Criteria:

1. Structural abnormalities of the nose or nasal polyposis, a history of frequent nosebleeds (more than once a month), nasal surgery (performed less than 12 months prior to signing the informed consent form), or ongoing upper respiratory tract infection.
2. Any respiratory disease, or any other acute infectious disease that has resolved less than 4 weeks prior to signing the informed consent form.
3. Any allergenspecific therapy (AIT) less than 3 years before signing the informed consent form.
4. Anaphylactic shock during AIT in the anamnesis.
5. Any immunopathological conditions and immunodeficiency.
6. Uncontrolled bronchial asthma that requires medical treatment.
7. Presence of clinically significant sensitization to year-round allergens (epidermal allergens, house dust allergens, etc.) at the time of screening.
8. Severe chronic or recurrent diseases that, according to the researcher, may interfere with AIT.
9. Convulsive seizures or a history of epilepsy.
10. Any chronic or recurrent infectious diseases in the anamnesis in the acute stage.
11. The presence of significant deviations according to physical examination, vital signs measurement, as well as laboratory tests, electrocardiography and fluorography / radiography of the lungs performed on analog (film) or digital fluorographs/X-ray machines, which in the opinion of the researcher may interfere with ASIT.
12. Malignancy of any nature and localization in the anamnesis.
13. A history of bone marrow transplantation (BMT) or peripheral blood hematopoietic stem cells (TSCC).
14. The presence of clinically significant cardiovascular and mental illnesses that, according to the researcher, may hinder the implementation of ASIT.
15. Dehydration due to diarrhea, vomiting, or other causes within 24 hours prior to subcutaneous injection of the test drug or placebo.
16. Blood donation or blood loss (450 ml of blood or more) less than 3 months before signing the informed consent.
17. Participation in clinical trials of any medications (less than 3 months or 5 half-lives from taking the study drug, whichever is longer) before subcutaneous administration of the study drug or placebo.
18. Regular alcohol consumption exceeding 5 units of alcohol per week or information about alcoholism, drug addiction, or drug abuse in the anamnesis.
19. Seropositive HIV status (presence of anti-HIV-1 and/or anti-HIV-2 in the blood) and/or detection of markers of acute hepatitis B (presence of HBsAg in the blood) and/or hepatitis C (presence of anti-HCV in the blood) and/or syphilis.
20. Surgery on ENT organs and/or any other surgical interventions planned for the period of participation in the study, except for those that can be performed on an outpatient basis and under local anesthesia (for example, tooth extraction, nevus removal, etc.).
21. The use of the following medications (the use of hormonal contraceptives is allowed):

    i. parenteral administration of steroid drugs within 12 weeks prior to signing of informed consent; ii. oral steroid medications within 8 weeks prior to signing informed consent; iii. inhaled and topical steroid medications within 4 weeks prior to signing the informed consent form; iv. beta-blockers, including topical forms, within 1 week prior to signing informed consent; v. MAO inhibitors in combination with sympathomimetics for 1 week prior to signing of informed consent; vi. vaccination with any vaccine within 4 weeks before signing the informed consent; vii. immunotherapy, including treatment with immunosuppressive or genetically engineered biological drugs (GBPS), within 24 weeks prior to signing the informed consent.
22. Pregnancy or breast-feeding.
23. Hypersensitivity to any of the components of the drug/placebo, with the exception of hypersensitivity to a causally significant allergen (birch pollen).
24. Psychological, family, sociological, or geographical conditions that potentially hinder compliance with the study protocol and follow-up schedule.
25. Unwillingness or inability to comply with the requirements of this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Daily Symptom Score (dSS) | Up to 3 months after the end of treatment.
  According to the dSS scale, the patient will need to assess the presence and severity of 4 symptoms of AR (itchy nose, sneezing, runny nose and nasal congestion) and 2 symptoms of AK (itchy eyes/redness of the eyes and lacrimation) on a 3-point scale, where 0 - no symptoms, 1-mild symptoms (the sign/symptom is clearly present, but causes minimal anxiety; easily tolerated), 2 - moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 - severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping).
  4 nasal and 2 conjunctival symptoms to be assessed from 0 to 3 score each. Total (dayli) symptoms score: 0-3 (max score is 3, i.e. 18 points/divided by 6 symptoms): 0 - no symptoms, 3 - severe symptoms.
Daily Medication Score (dMS) | Up to 3 months after the end of treatment.
  The use of the following medications that can be used to relieve symptoms of allergic rhinitis and allergic conjunctivitis will need to be evaluated by the patient
  * Non-sedative H1-antihistamines (H1A) for oral and / or topical use (eyes or nose) = 1 point;
  * Intranasal corticosteroids (InCS) with / without H1A = 2 points;
  * Oral corticosteroids with / without InKS, with / without H1A = 3 points. Points are not added up, and the maximum score is set. Thus, the minimum dMS value is 0 and means no need for medication, and the maximum dMS value is 3 and means the need for third-line medications).
Combined Symptom and Medication Score (CSMS) | Up to 3 months after the end of treatment.
  The eDP automatically calculates total dSS and dMS scores based on the patient's daily scores:
  * The (Total) Daily Symptoms Score (dSS) is the sum of the scores for each of the symptoms and can range from 0 to 3 points
  * The (Total) Daily Medication Score (dMS): 0-3 (max score is 3)
  СSMS= dSS (0-3) + dMS (0-3) CSMS can range from 0 to 6 points, where the minimum value is 0 points and means no symptoms and no need for medication, and the maximum value is 6 points and means the maximum severity of rhinitis symptoms, despite the use of third-line medications.

SECONDARY OUTCOMES:
36-Item Short Form Health Survey (36-SF) | Day 0, week 16 (end of treatment) and up to 3 months after the end of treatment.
  The questionnaire reflects the overall well-being and degree of satisfaction with those aspects of a person's life that are affected by the state of health.
  The SF-36 consists of 36 questions, grouped into eight scales: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The scores for each scale are constructed so that a higher value (from 0 to 100) indicates a more favorable health state for that particular scale.
Severity of allergic rhinitis symptoms on a Visual-analog scale (VAS) | Uo to 3 months after the end of therapy.
  VAS is a horizontal graded line 10 cm long on which the patient marks with a vertical line the assessment of the effect of AR on their well - being, expressed in points from 0 to 100 (from 0 to 10 cm), where 0 is the absence of complaints and symptoms, and 100 is the most pronounced manifestations of the disease. Results from 0 to 50 points (5 cm) indicate a controlled course of allergic AR, from 50 points and above (≥5 cm) - an uncontrolled course of AR.
Antibody level to the Betv1, Mald1 and PreS antigens. | Day 1, week 8, week 16 and up to 3 months after the end of treatment.
  IgG, IgE, IgA, IgM antibody level to all three antigen will be assessed.
Percentage of the CD3+CD69+ T-cells | Day 1, week 8, week 16 and up to 3 months after the end of treatment.
  Assessment of CD3+CD69+ - percentage of cells expressing the marker and geometric mean fluorescence intensity in peripheral blood cells without in vitro activation.
Cytokines level | Day 1, week 8, week 16 and up th 3 months after the end of treatment.
  Cytokins level: IL-1β, IFNγ, IL-2, IL-4, IL-5, IL-10, IL-13 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair
Locations (1):
- National Research Center - Institute of Immunology Federal Medical-Biological Agency, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No